## A PROSPECTIVE RANDOMIZED STUDY COMPARING THE INCIDENCE OF RADIAL ARTERY OCCLUSION (RAO) AND THE TIME TO HEMOSTASIS (TTH) WHEN USING A HEMOSTASIS BAND ALONE AND IN CONJUNCTION WITH A DISC COMPRISED OF POTASSIUM FERRATE (STATSEAL ADVANCED) FOLLOWING TRANSRADIAL CATHETERIZATION. Study Sponsor: A Physician Initiated Study

Principal Investigator: Arnold Seto, MD, MPA

Cardiology Division Veterans Medical Center Long Beach

## Statistical Analysis

Continuous data are presented as mean ± standard deviation and as median [interquartile range], and compared using unpaired t-test and Mann-Whitney U-test, respectively. Discrete data are presented as frequencies with their respective percentages and compared using Fisher's exact test. Outcome data were analyzed on an intention-to-treat basis. Two-tailed tests of significance are reported and p values < 0.05 were considered statistically significant. Univariate logistic regression was performed using all baseline patient and procedural variables available to predict the secondary outcome of hematoma formation. Variables that were significant in univariate analysis at p<0.25 were retained and entered into a multivariate model with a threshold of p<0.05 being considered as significant. Statistical analyses were performed using the SPSS statistical software program (SPSS version 16.0.2, Chicago, IL).